CLINICAL TRIAL: NCT04433507
Title: Antireflux Efficacy of Hiatal Hernia Repairs Concomitant to Sleeve Gastrectomy in Obese Patients (BMI 35-50)
Brief Title: Antireflux Efficacy of Hiatal Hernia Repairs in Sleeve Gastrectomy Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Radu Pescarus, Principal Investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CER-2019-1642
Record Dates: First submitted 2019-06-07; First posted 2020-06-16 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Gastroesophageal Reflux
Keywords: Sleeve Gastrectomy; Gastroesophageal reflux; Bariatric Surgery; Complications
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: 50 patients in the SG group and 50 in the SG + primary hiatal hernia repair group following randomization
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeve Gastrectomy group (Active Comparator): This group will receive a Sleeve Gastrectomy only, a mainly restrictive procedure which consists in creating a narrow tube-like stomach based on its lesser curvature.
  Interventions: Procedure: Sleeve gastrectomy
- Sleeve Gastrectomy + Hiatal Hernia repair group (Experimental): This group will receive a Sleeve Gastrectomy combined with hiatal hernia repair. Hiatal Hernia repair consists of a peri-esophageal dissection proximal to the diaphragmatic crura to achieve an intra-abdominal esophageal length of 2-3 cm. The pillars will then be closed anteriorly and posteriorly using nonabsorbable sutures.
  Interventions: Procedure: Sleeve gastrectomy; Procedure: Hiatal Hernia repair

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Laparoscopic sleeve gastrectomy (LSG) is performed through a standard 5-port technique. After dissection of the greater curvature of the stomach, a narrow tube-like stomach is created after stapling off the lateral aspect of the stomach using a 40 French bougie as a guide.
Procedure: Hiatal Hernia repair — Hiatal hernia repair consists in a circumferential dissection of the diaphragmatic crura to achieve an intra abdominal esophageal length of 2-3 cm. The crura will then be closed anteriorly and posteriorly using nonabsorbable sutures.
  Arms: Sleeve Gastrectomy + Hiatal Hernia repair group

SUMMARY:
Gastroesophageal reflux (GR) occurrence or persistence following a sleeve gastrectomy (SG) can be correlated to several factors but it is clear that one of the key factors is a persistent hiatal hernia or laxity of the esophageal hiatus. However, there are no clear guidelines presently available on surgical management of small size hernias or an abnormal hiatus. Therefore, hiatal hernia management is decided intraoperatively by the operating surgeon. The main goal of this study is to evaluate the efficacy of primary hiatal hernia repairs on gastroesophageal reflux concomitant to sleeve gastrectomy. The secondary objectives are hiatal hernia recurrence following primary surgery and the occurrence of "de novo" GR.

DETAILED DESCRIPTION:
Background :

The Sleeve gastrectomy (SG) is the most common bariatric procedure worldwide because it is the simplest to perform, from a technical standpoint, and the most efficient in terms of metabolic control and weight loss. However, this intervention can lead to several complications, including the onset or intensification of gastroesophageal reflux (GR) with the associated impact on the patients' quality of life and a possible evolution into Barrett's esophagus. One of the key factors in the development of this complication is a persistent hiatal hernia.

Aims: The main objective of this study is to provide an objective evaluation of the effect of primary hiatal hernia repair on GR concomitant to sleeve gastrectomy. The secondary objectives are hiatal hernia recurrence following primary surgery and the occurrence of "de novo" GR.

Methods :

A total of 100 patients will be recruited for the pilot study, with 50 patients in the SG group and 50 in the SG + primary hiatal hernia repair group following randomization. Then, based on a sample size study, recruitment will be continued as needed. None of the procedures performed are experimental. All obese patients with a BMI between 35-50, aged 18-65 and undergoing surgery for a SG in the institution's bariatric surgery department will be eligible to participate in this study. Exclusion criteria will be hiatal hernias greater than 2 cm, a hiatal repair requiring a drain, prior bariatric surgery or any other counterindication to SG. All patients will be evaluated preoperatively using: 1) EGD, 2) esophageal manometric study, 3) pH assessment and 4) validated GR questionnaires (GERD-HRPL; GCSI). Iconographic intraoperative data on hiatal morphology and the type of cure used will be collected and records will be kept according to Ethics committee guidelines. After a 6-month follow-up the participants will undergo the same tests, including questionnaires, for a medium-term profile.

ELIGIBILITY:
Inclusion Criteria:

* All obese patients with a BMI between 35-50
* Aged 18-65 and undergoing surgery for a Sleeve Gastrectomy in institution's bariatric surgery department

Exclusion Criteria:

* hiatal hernias greater than 2 cm,
* hiatal repair requiring mesh placement
* prior bariatric surgery or any other counterindication to Sleeve Gastrectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in the presence of pathological Gastroesophageal reflux disease (GERD) | Before surgery and 6 months after surgery
  Pathological GERD will be assessed objectively using a 24 hour pH study and an EGD (esophagogastroduodenoscopy - presence of esophagitis)

SECONDARY OUTCOMES:
Presence of hiatal hernia (intrathoracic migration of the sleeve) | Before surgery and 6 months postoperative
  Presence of hiatal hernia will be assessed using EGD and high-resolution esophageal manometry
Presence of hypotensive lower esophageal sphincter (LES) | before the surgery and 6 months post-operative
  Hypotensive LES will be measured objectively using a high-resolution esophageal manometry study
Worsening or new-onset gastroesophageal reflux disease | before the surgery and 6 months post-operative
  Worsening or new-onset gastroesophageal reflux disease will be measured using a validated reflux questionnaire (GERD-HRQL). The GERD-HRQL questionnaire was developed and validated to measure changes of typical GERD symptoms such as heartburn and regurgitation in response to surgical or medical treatment. Total Score: Calculated by summing the individual scores to questions 1-15.
  Greatest possible score (worst symptoms) = 75 Lowest possible score (no symptoms) = 0

CONTACTS AND LOCATIONS:
Overall Officials: Radu Pescarus, MD, Principal Investigator — Hopital Sacré Coeur de Montréal
Locations (1):
- Hopital Sacré-Coeur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No